CLINICAL TRIAL: NCT02508480
Title: Testing Effectiveness of a Peer-Led Intervention to Enhance Community Integration
Acronym: Photovoice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Zlatka Russinova, Research Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2014-22
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Mental Disorders
Keywords: Stigma; Community Integration
MeSH Terms: conditions — Mental Disorders; Social Stigma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Photovoice (Experimental): Participants in this arm will attend a 10-week peer-led Photovoice program conducted in group format.
  Interventions: Behavioral: Photovoice
- Enhanced Control (Active Comparator): Participants in this arm will attend a 60-minute peer-led group discussion on stigma and discrimination, and be eligible to participate in the 10-week Photovoice program after completing all study assessments.
  Interventions: Behavioral: Enhanced Control

INTERVENTIONS:
Behavioral: Photovoice — The 10-session, peer-led Photovoice program, designed to empower individuals with SMI to confront public prejudice and discrimination and reduce personal stigma (self-stigma and perceived stigma), was developed and pilot tested at our Center, with primary contributions from staff with a lived experience of mental illness.
  In the Photovoice sessions, participants will be given a workbook titled Combating Prejudice and Discrimination through Photovoice Empowerment. Peer leaders will facilitate discussions based on topics in the workbook. Participants will be given cameras and guidance on taking pictures and writing narratives descriptions about the pictures, specifically the ways in which the pictures relate to experiences of prejudice and discrimination.
  Arms: Photovoice
Behavioral: Enhanced Control — The control SAU condition will be enhanced with a 60-minute peer-led manualized educational group session (Leaders' Guidelines and Handout for Participants are attached). It will provide participants with information about the nature of stigma and the laws in the U.S. that protect people with disabilities from discrimination. Participants will be engaged in a discussion about their use of different strategies for proactive coping with psychiatric stigma. This session will be co-led by the same peers who will be delivering the Photovoice program to the experimental group at relevant wave and study sites. Participants randomized to the enhanced Services as Usual control condition will be invited to join a Photovoice group once they complete the final 6-month follow-up assessment.
  Arms: Enhanced Control

SUMMARY:
We are conducting a randomized clinical trial (RCT) comparing the 10-week peer-led Photovoice program to services as usual (SAU) at a large publicly funded community mental health agency in Massachusetts. The control SAU condition will be enhanced with a 60-minute peer-led group educational session about understanding and coping with prejudice and discrimination. The 10-session, peer-led Photovoice program, designed to empower individuals with serious mental illness (SMI) to confront public prejudice and discrimination and reduce personal stigma (self-stigma and perceived stigma), was developed and pilot tested at our Center, with primary contributions from staff with a lived experience of mental illness. Development of the Photovoice program was guided by an adaptation of the stress-coping model, informed by recent research and conceptualizations of the effects of stigma on people with SMI. The stress-coping model explicates the mechanisms by which public stigma about mental illness can lead to personal stigma, which in turn has a negative impact on the person's mental health and psychosocial functioning. This model also identifies critical factors that contribute to personal stigma or protect against it, as well as more vs. less adaptive coping responses, that are the primary focus of the Photovoice program.

DETAILED DESCRIPTION:
We are conducting a RCT comparing the 10-week peer-led Photovoice program to services as usual (SAU) enhanced with a 60-minute peer-led group discussion session. The RCT will be at a large publicly funded community mental health agency in Massachusetts. A total of 192 participants or 96 participants per group will be recruited over a period of 36 months across the three clubhouses of the agency where the intervention will take place. We plan to have randomization cohorts of 16 individuals per delivery of the Photovoice program at each of the three clubhouses. Given the projected sample size of 192 participants, we will have 12 randomization cohorts - 4 at each clubhouse implemented at 6-month intervals. Participants will be randomized to either the Photovoice program (plus usual services) or the enhanced SAU. Participants will be assessed by a blinded rater at baseline, post-treatment, 3-month and 6-month follow-ups on a range of primary and secondary outcomes related to personal stigma, coping, and functioning. Primary analyses will test the hypotheses that the Photovoice program will lead to significantly greater reductions in self-stigma and perceived stigma, greater improvements in proactive coping with psychiatric prejudice and discrimination, and greater improvements in community functioning and integration than the enhanced SAU. Secondary analyses will evaluate whether the Photovoice program leads to greater gains than SAU in psychological adjustment, including wellbeing, personal growth and recovery. Individuals randomized to the enhanced SAU will be able to join the 10-week Photovoice program once they complete their 6-month follow up for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18years and older
* Diagnosis of serious mental illness
* Receiving services at agency where study is taking place
* Willing and able to give written consent
* Conversant in English

Exclusion Criteria:

* Prior exposure to Photovoice
* Cognitive disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zlatka Russinova, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Photovoice: Participants in this arm will attend a 10-week peer-led Photovoice program conducted in group format.
  Photovoice: The 10-session, peer-led Photovoice program, designed to empower individuals with SMI to confront public prejudice and discrimination and reduce personal stigma (self-stigma and perceived stigma), was developed and pilot tested at our Center, with primary contributions from staff with a lived experience of mental illness.
  In the Photovoice sessions, participants will be given a workbook titled Combating Prejudice and Discrimination through Photovoice Empowerment. Peer leaders will facilitate discussions based on topics in the workbook. Participants will be given cameras and guidance on taking pictures and writing narratives descriptions about the pictures, specifically the ways in which the pictures relate to experiences of prejudice and discrimination.
- Enhanced Control: Participants in this arm will attend a 60-minute peer-led group discussion on stigma and discrimination, and be eligible to participate in the 10-week Photovoice program after completing all study assessments.
  Enhanced Control: The control SAU condition will be enhanced with a 60-minute peer-led manualized educational group session. It will provide participants with information about the nature of stigma and the laws in the U.S. that protect people with disabilities from discrimination. Participants will be engaged in a discussion about their use of different strategies for proactive coping with psychiatric stigma. This session will be co-led by the same peers who will be delivering the Photovoice program to the experimental group at relevant wave and study sites. Participants randomized to the enhanced Services as Usual control condition will be invited to join a Photovoice group once they complete the final 6-month fo
Period: Overall Study
Arm/Group | Photovoice | Enhanced Control
Started | 95 | 97
Post-Treatment Assessment (Participants who completed assessment after the 10-week photovoice intervention) | 87 | 89
Three Month Follow-up (Participants who completed the 3-month post-intervention follow-up) | 84 | 86
Six-Month Follow-Up (Participants who completed the 6-month post-intervention follow-up) | 84 | 86
Completed (Participants who completed at least one post-baseline assessment over the study period.) | 90 | 93
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Photovoice | Enhanced Control | Total
Number analyzed (Participants) | 95 | 97 | 192
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.36 (13.37) | 47.48 (13.86) | 46.93 (13.60)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 54 | 50 | 104
  Female | 40 | 46 | 86
  Other | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 84 | 82 | 166
  Black | 3 | 7 | 10
  Asian | 1 | 0 | 1
  White, hispanic | 2 | 2 | 4
  Multi-racial/ Other | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 95 | 97 | 192

OUTCOME MEASURES:

1. Primary Outcome: Internalized Stigma of Mental Illness Scale, Change in Internalized Stigma
Description: a 29-item, 4-point scale (strongly disagree to strongly agree) assesses behaviors, thoughts and feelings that are self-stigmatizing and includes alienation, stereotype endorsement, discriminatory experiences, social withdrawal, and stigma resistance subscales. Internal consistency is .9 and test-retest reliability is .92. Lower scores are better.
  The scale score is the average score on the 29 items, which are scored from 1-4. Lower scores signify less internalized stigma.
Time Frame: Baseline, post-treatment, 3 months post-treatment, 6 months post-treatment
Population: Participants included in analysis at each time point are those who completed the scale at that time point.
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Photovoice | Enhanced Control
Number analyzed (Participants) | 95 | 97
Score on a scale.
  Baseline | 2.18 (0.40) | 2.09 (0.42)
  Post-Intervention: number analyzed (Participants) | 87 | 88
  Post-Intervention | 2.11 (0.40) | 2.05 (0.45)
  3-Month follow-up: number analyzed (Participants) | 84 | 86
  3-Month follow-up | 2.64 (0.37) | 2.71 (0.31)
  6-Month follow-up: number analyzed (Participants) | 84 | 89
  6-Month follow-up | 2.08 (0.41) | 2.01 (0.43)
Statistical Analysis 1: Comparison: Photovoice vs Enhanced Control; The two study arms were compared using mixed models analysis controlling for baseline scores. Variables included in the model were- baseline score, group, time, and group by time interaction. The p-value reported below is for group effect; Test type: Superiority; p = 0.66, Mixed Models Analysis

2. Primary Outcome: Approaches to Coping With Stigma, Change in Coping With Stigma
Description: is a 27-item, 4-point scale ranging from 1-4 (strongly disagree to strongly agree) measuring strategies to cope with stigma: secrecy, withdrawal, distancing, educating others, and challenging others. The average score of the items in the first three subscales will represent the index for Avoidant Coping and the average score of the items in the last two subscales - the index for Proactive Coping with Stigma. Internal consistency for subscales range: .63-.84. Lower scores are better on Avoidant Coping and higher scores are better on Proactive Coping.
Time Frame: Baseline, post-treatment, 3 months post-treatment, 6 months post-treatment
Population: Participants included in analysis at each time point are those who completed the scale at that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photovoice | Enhanced Control
Number analyzed (Participants) | 95 | 97
score on a scale
  Proactive Coping- Baseline | 2.90 (0.42) | 2.93 (0.47)
  Proactive Coping- Post-Intervention: number analyzed (Participants) | 87 | 88
  Proactive Coping- Post-Intervention | 2.87 (0.39) | 2.97 (0.47)
  Proactive Coping- 3-Month follow-up: number analyzed (Participants) | 84 | 86
  Proactive Coping- 3-Month follow-up | 2.06 (0.49) | 1.87 (0.43)
  Proactive Coping- 6-Month follow-up: number analyzed (Participants) | 84 | 89
  Proactive Coping- 6-Month follow-up | 2.86 (0.48) | 2.96 (0.56)
  Avoidant Coping- Baseline | 2.53 (0.33) | 2.51 (0.30)
  Avoidant Coping- Post-Intervention: number analyzed (Participants) | 87 | 88
  Avoidant Coping- Post-Intervention | 2.52 (0.32) | 2.46 (0.38)
  Avoidant Coping- 3-Month Follow-Up: number analyzed (Participants) | 84 | 86
  Avoidant Coping- 3-Month Follow-Up | 2.41 (0.44) | 2.31 (0.56)
  Avoidant Coping- 6-Month Follow-Up: number analyzed (Participants) | 84 | 89
  Avoidant Coping- 6-Month Follow-Up | 2.52 (0.36) | 2.45 (0.35)
Statistical Analysis 1: Comparison: Photovoice vs Enhanced Control; The two study arms were compared using mixed models analysis controlling for baseline scores. Variables included in the model were- baseline score, group, time, and group by time interaction. The p-value reported below is for group effect for Proactive Coping; Test type: Superiority; p = 0.884, Mixed Models Analysis — Group effect for Proactive Coping
Statistical Analysis 2: Comparison: Photovoice vs Enhanced Control; The two study arms were compared using mixed models analysis controlling for baseline scores. Variables included in the model were- baseline score, group, time, and group by time interaction. The p-value reported below is for group effect for Avoidant Coping; Test type: Superiority; p = 0.543, Mixed Models Analysis — Group effect for Avoidant Coping

3. Primary Outcome: The Stigma Scale, Change in Perceptions of Stigma
Description: is a 28 item, 5 point scale ranging from 0-4 (strongly disagree to strongly agree) measuring experienced and anticipated stigma. Internal consistency ranges from .85-.87 and test-retest reliability from .4 to .7. The scale score is the average score on all items. Lower scores are better.
Time Frame: Baseline, post-treatment, 3 months post-treatment, 6 months post-treatment
Population: Participants included in the analysis at each time point are those who completed the scale at that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photovoice | Enhanced Control
Number analyzed (Participants) | 95 | 97
score on a scale
  Baseline | 1.92 (0.59) | 1.81 (0.61)
  Post-Intervention: number analyzed (Participants) | 87 | 88
  Post-Intervention | 1.87 (0.59) | 1.75 (0.66)
  3-Month follow-up: number analyzed (Participants) | 84 | 86
  3-Month follow-up | 1.87 (0.56) | 1.82 (0.64)
  6-Month follow-up: number analyzed (Participants) | 84 | 89
  6-Month follow-up | 1.78 (0.60) | 1.76 (0.63)
Statistical Analysis 1: Comparison: Photovoice vs Enhanced Control; The two study arms were compared using mixed models analysis controlling for baseline scores. Variables included in the model were- baseline score, group, time, and group by time interaction; Test type: Superiority; p = 0.135, Mixed Models Analysis — The p-value above is for the overall group effect

4. Primary Outcome: Heinrich's Quality of Life Scale-Client Version, Change in Quality of Life
Description: This is a 21 item, semi-structured interview-based, rating of an individual's psycho-social functioning and satisfaction with various life domains. The score on each item ranges from 0-6 with higher scores indicating better functioning. The subscale scores are computed based on the average score of items included.
  We report below on the interpersonal functioning and intrapsychic foundations subscales.
Time Frame: Baseline, post-treatment, 3 months post-treatment, 6 months post-treatment
Population: Participants included in the analysis at each time point are participants who completed the measure at that time point.
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Photovoice | Enhanced Control
Number analyzed (Participants) | 95 | 97
Score on a scale.
  Baseline-Interpersonal | 2.79 (1.06) | 2.94 (1.08)
  Post-Intervention-Interpersonal: number analyzed (Participants) | 87 | 89
  Post-Intervention-Interpersonal | 2.82 (1.03) | 3.10 (1.13)
  3-Month follow-up-Interpersonal: number analyzed (Participants) | 83 | 86
  3-Month follow-up-Interpersonal | 2.86 (1.09) | 2.98 (1.09)
  6-Month follow-up-Interpersonal: number analyzed (Participants) | 83 | 89
  6-Month follow-up-Interpersonal | 2.98 (0.99) | 3.11 (1.03)
  Baseline- Intrapsychic | 3.35 (0.96) | 3.61 (0.97)
  Post-intervention- Intrapsychic: number analyzed (Participants) | 87 | 89
  Post-intervention- Intrapsychic | 3.43 (0.97) | 3.42 (0.91)
  3-Month follow-up- Intrapsychic: number analyzed (Participants) | 83 | 86
  3-Month follow-up- Intrapsychic | 3.34 (1.04) | 3.34 (0.91)
  6-Month follow-up- Intrapsychic: number analyzed (Participants) | 83 | 89
  6-Month follow-up- Intrapsychic | 3.37 (0.95) | 3.39 (0.87)
Statistical Analysis 1: Comparison: Photovoice vs Enhanced Control; The two study arms were compared on the interpersonal function subscale using mixed models analysis controlling for baseline scores. Variables included in the model were- baseline score, group, time, and group by time interaction; Test type: Superiority; p = 0.25, Mixed Models Analysis — The p-value above represents the overall group effect
Statistical Analysis 2: Comparison: Photovoice vs Enhanced Control; The two study arms were compared on the intrapsychic foundations subscale using mixed models analysis controlling for baseline scores. Variables included in the model were- baseline score, group, time, and group by time interaction; Test type: Superiority; p = 0.118, Mixed Models Analysis — The p-value represents the overall group effect

5. Primary Outcome: Temple University Community Participation Scale, Change in Community Participation
Description: is a 26 item instrument measuring frequency of participation and importance of various community activities (e.g., movies, library). Test-retest reliability is .7 and internal consistency is .9. Higher scores are better.
  We provide below the results for cumulative days of participation in the last 30 days across the 26 activities included in the measure (tcpm_days_participated). The possible range for this measure is 0-780.
Time Frame: Baseline, post-treatment, 3 months post-treatment, 6 months post-treatment
Population: Participants included in the analysis at each time point are those who completed the questionnaire at that time point.
Measure: Mean (Standard Deviation); unit: Days of participation
Arm/Group | Photovoice | Enhanced Control
Number analyzed (Participants) | 95 | 97
Days of participation
  tcpm_days_participated- Baseline | 51.25 (31.74) | 54.80 (34.74)
  tcpm_days_participated-Post-Intervention: number analyzed (Participants) | 87 | 89
  tcpm_days_participated-Post-Intervention | 47.40 (26.81) | 48.99 (33.96)
  tcpm_days_participated-3-Month follow-up: number analyzed (Participants) | 84 | 86
  tcpm_days_participated-3-Month follow-up | 45.75 (29.56) | 47.76 (30.90)
  tcpm_days_participated-6-Month follow-up: number analyzed (Participants) | 84 | 89
  tcpm_days_participated-6-Month follow-up | 45.10 (26.93) | 44.17 (29.11)
Statistical Analysis 1: Comparison: Photovoice vs Enhanced Control; The two study arms were compared using mixed models analysis controlling for baseline scores. Variables included in the model were- baseline score, group, time, and group by time interaction. The p-value reported below is for group effect for tcpm_days_participated; Test type: Superiority; p = 0.917, Mixed Models Analysis — The p-value is for group effect for tcpm_days_participated

6. Secondary Outcome: Brief Psychiatric Rating Scale, Change in Psychiatric Symptoms
Description: This is a 24-item scale that rates the severity of a variety of psychiatric psychotic symptoms, positive and negative symptoms on a 7-point scale of 1 (absent) to 7 (severe). The scale score is the mean of the score on all items, ranging from 1 to 7.
Time Frame: Baseline, post-treatment, 3 months post-treatment, 6 months post-treatment
Population: The number analyzed at each time point represent the number who completed the assessment at that time point.
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Photovoice | Enhanced Control
Number analyzed (Participants) | 95 | 97
Score on a scale.
  Baseline | 1.79 (0.47) | 1.78 (0.41)
  Post-Intervention: number analyzed (Participants) | 87 | 88
  Post-Intervention | 1.71 (0.43) | 1.80 (0.43)
  3-Month follow-up: number analyzed (Participants) | 83 | 86
  3-Month follow-up | 1.77 (0.42) | 1.85 (0.43)
  6-Month follow-up: number analyzed (Participants) | 83 | 88
  6-Month follow-up | 1.78 (0.45) | 1.72 (0.39)
Statistical Analysis 1: Comparison: Photovoice vs Enhanced Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.017, Mixed Models Analysis — The p-value above is for the overall group effect

7. Secondary Outcome: Scales of Psychological Well-Being, Change in Well-being
Description: This is a 54-item, 6-point (1 to 6) measure rating wellbeing (from strongly disagree to strongly agree) including subscales of mastery, personal growth, purpose in life, self-acceptance, autonomy and positive relations with others. Internal consistency is .94. It has been successfully used with individuals with SMI. Higher scores indicate greater well-being.
  Each subscale score is the average of the scores on included items. We present below the scores on the self-acceptance subscale.
Time Frame: Baseline, post-treatment, 3 months post-treatment, 6 months post-treatment
Population: The participants included in analysis at each time point are those who completed the measure at that time point.
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Photovoice | Enhanced Control
Number analyzed (Participants) | 95 | 97
Score on a scale.
  Baseline | 3.75 (1.02) | 3.92 (1.07)
  Post-Intervention: number analyzed (Participants) | 87 | 88
  Post-Intervention | 3.83 (1.06) | 3.90 (0.95)
  3-Month follow-up: number analyzed (Participants) | 84 | 86
  3-Month follow-up | 3.86 (0.95) | 3.81 (1.04)
  6-Month follow-up: number analyzed (Participants) | 84 | 88
  6-Month follow-up | 3.96 (1.07) | 3.89 (0.96)
Statistical Analysis 1: Comparison: Photovoice vs Enhanced Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.597, Mixed Models Analysis — The p-value above represents the overall group effect

8. Secondary Outcome: Maryland Assessment of Recovery, Change in Perceptions of Recovery
Description: is a 25-item, 5-point (1 to 5) scale that assesses a person's sense of recovery from mental illness across a variety of dimensions. Internal consistency is.95 and test-retest reliability is .89). The scale score is the average score on each item with higher scores indicating higher levels of recovery.
Time Frame: Baseline, post-treatment, 3 months post-treatment, 6 months post-treatment
Population: Participants included in the analysis at each time point are those who completed the measure at that timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Photovoice | Enhanced Control
Number analyzed (Participants) | 95 | 97
Score on a scale.
  Baseline | 3.95 (0.43) | 4.07 (0.51)
  Post-Intervention: number analyzed (Participants) | 87 | 88
  Post-Intervention | 3.94 (0.54) | 4.07 (0.54)
  3-Month follow-up: number analyzed (Participants) | 84 | 86
  3-Month follow-up | 3.92 (0.53) | 4.05 (0.48)
  6-Month follow-up: number analyzed (Participants) | 84 | 89
  6-Month follow-up | 4.02 (0.55) | 4.02 (0.52)
Statistical Analysis 1: Comparison: Photovoice vs Enhanced Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.076, Mixed Models Analysis — The p-value above represents the overall group effect

9. Secondary Outcome: Personal Growth and Recovery Scale, Change in Perceptions of Growth and Recovery
Description: This is a 16-item, 4 point scale (1 to 4) developed for a previous Photovoice study. Items tap aspects of a person's psychosocial functioning and recovery. Internal consistency is 0.94 and retest reliability is .79. The scale score is the average of scores on each item with higher scores indicating higher levels of recovery.
Time Frame: Baseline, post-treatment, 3 months post-treatment, 6 months post-treatment
Population: The participants included in analysis at each time point are those who completed the measure at that time point.
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Photovoice | Enhanced Control
Number analyzed (Participants) | 95 | 97
Score on a scale.
  Baseline | 3.31 (0.58) | 3.38 (0.57)
  Post-Intervention: number analyzed (Participants) | 87 | 88
  Post-Intervention | 3.31 (0.61) | 3.36 (0.56)
  3-Month follow-up: number analyzed (Participants) | 84 | 86
  3-Month follow-up | 3.32 (0.6) | 3.36 (0.58)
  6-Month follow-up: number analyzed (Participants) | 84 | 89
  6-Month follow-up | 3.38 (0.57) | 3.43 (0.55)
Statistical Analysis 1: Comparison: Photovoice vs Enhanced Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.978, Mixed Models Analysis — The p-value above represents the overall group effect

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of study participation for each individual enrolled, which was 9 months.
Arm/Group | Photovoice | Enhanced Control
All-Cause Mortality (participants affected / at risk) | 1/95 | 2/97
Serious Adverse Events (participants affected / at risk) | 1/95 | 2/97
Other Adverse Events (participants affected / at risk) | 0/95 | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photovoice (N=95) | Enhanced Control (N=97)
Death (General disorders) | 1 (1) | 2 (2) — Participant death due to existing medical conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT02508480/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT02508480/SAP_001.pdf